CLINICAL TRIAL: NCT00603317
Title: Pharmacodynamic Drug Interaction Between Warfarin and Amoxicillin-clavulanic Acid
Acronym: INWARA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Valerie MILLUL, Department Clinical Reseach of Developpement
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P051056
Record Dates: First submitted 2008-01-16; First posted 2008-01-29 (Estimated); Last update posted 2010-07-12 (Estimated); Status verified 2010-05

CONDITIONS: Oral Anticoagulation; Deep Venous Thrombosis; Atrial Fibrillation; Pulmonary Embolism
Keywords: Warfarin; Drug interaction; Pharmacogenetics; Amoxicillin; Clavulanic acid
MeSH Terms: conditions — Venous Thrombosis; Atrial Fibrillation; Pulmonary Embolism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Order 1 : Firstly Amoxicillin-Acid clavulanic, and Secondly Placebo
  Interventions: Drug: Firstly : Amoxicillin-Clavulanic acid and secondly : Placebo
- 2 (Experimental): Order 2 : Firstly Placebo, and Secondly Amoxicillin-Acid clavulanic
  Interventions: Drug: Firstly : Placebo and secondly : Amoxicillin-Clavulanic acid

INTERVENTIONS:
Drug: Firstly : Amoxicillin-Clavulanic acid and secondly : Placebo — Amoxicillin : 2g twice daily Clavulanic acid : 125 mg twice daily
  Arms: 1
Drug: Firstly : Placebo and secondly : Amoxicillin-Clavulanic acid — Amoxicillin : 2g twice daily Clavulanic acid : 125mg twice daily seven consecutive days
  Arms: 2

SUMMARY:
Several case reports indicate that the use of the antibiotic combination amoxicillin and clavulanic acid (AM-CLAVAC) can interact with warfarin pharmacodynamics. However, fever per se might also be responsible of these warfarin overdose reports, as well as the use of high dose paracetamol.

The aim of the present study is to determine if AM-CLAVAC can increase the pharmacodynamics of warfarin among patients at steady state Double blinded cross over controlled study vs placebo performed in 12 evaluable patients treated with warfarin with an INR target 2 to 3 and a stable INR and a stable dose.

DETAILED DESCRIPTION:
Double blinded cross over controlled study vs placebo performed in 12 evaluable patients treated with warfarin with an INR target 2 to 3 and a stable INR and a stable dose

One period : seven consecutive days of amoxicillin(2g twice daily)- clavulanic acid (125 mg twice daily) association Wash out period of at least 4 weak with the return to a stable INR and warfarin dose One period : seven consecutive days of placebo twice daily

Main outcome INR delta Day7-Day

ELIGIBILITY:
Inclusion Criteria:

* patients treated with warfarin (target INR 2 to 3)
* stable anticoagulation (3 consecutive INR in the target)
* stable dose
* no infection
* normal CRP
* age >18 years
* normal transaminase levels

Exclusion Criteria:

* drug allergy
* penicillin allergy
* Alzheimer
* cancer
* thyroid disease
* gastro intestinal chronic disease
* frequent nausea or vomiting
* Cirrhosis
* chronic renal failure (GFR<60 ml/min)
* frequent intake of paracetamol or NSAID
* addict to drugs or alcool
* St John's wort treatment or grapefruit juice intake
* concomitant drugs (amiodarone, cimetidine, SSRI, clofibrate, fenofibrate, diltiazem, fluconazole, itraconazole, isoniazide, voriconazole, métronidazole, miconazole , omeprazole, glucocorticoids, zileuton, ritonavir, rifampicin, carbamazepine, phenytoin, phenobarbital)
* antibiotic use during the 3 last weeks
* pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
INR at day one and seven (delta Day7-Day1) | 7 days

SECONDARY OUTCOMES:
% of patients with an INR>3.5 during each study period mean INR during each study period effect of VKORC1 genetic polymorphism trough blood concentrations of S and R warfarin at day1 and day7 (delta) during each study period | 7 days for each period

CONTACTS AND LOCATIONS:
Overall Officials: Stephane MD MOULY, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital Lariboisière - Service de médecine interne, Paris, France